CLINICAL TRIAL: NCT06830265
Title: Comparing a Standard of Care Prostate Biopsy System with a Novel System Using Standard As Well As Computational Pathology Analyses to Measure Clinical and Morphometric Parameters.
Brief Title: Comparing Standard of Care Biopsy System to a Novel Biopsy Needle System by Computational Pathologic Analysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uro-1 Medical (Industry)
Collaborators: Duke University (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 25-001
Record Dates: First submitted 2025-01-22; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer Screening

STUDY DESIGN:
Intervention Model Description: Each patient enrolled will have prostate biopsy completed with a standard of care needle biopsy system (control) and a novel needle biopsy system (test), each targeting separate regions of the prostate.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test group (Active Comparator): The prostate of each subject will have a tissue removed by one needle in one lobe and the other needle in the other lobe.
  Interventions: Device: Novel needle biopsy catheter (test)
- Single Arm (Active Comparator): The prostate will be biopsied in one lobe by the control needle biopsy system and the other lobe by the test needle biopsy system.
  Interventions: Device: Novel needle biopsy catheter (test)

INTERVENTIONS:
Device: Novel needle biopsy catheter (test) — Tissue is collected from the prostate by introducing a needle into the prostate and cutting out a sample

SUMMARY:
Prostate biopsy is the definitive examination to establish the diagnosis of prostate cancer, but up to 40% of these biopsies overestimate or underestimate the severity of the disease. A novel biopsy needle system captures substantially more tissue than standard of care needles, but it is important to assess the retrieval of tissue for pathologic analyses. This study will compare quality and quantity of tissue retrieved by both systems. Further, tissue will be analyzed using computational pathology algorithms for atypical small acinar proliferation and Gleason scores in terms of tissue area, tissue length, and tissue tortuosity.

DETAILED DESCRIPTION:
Prostate tissue captured in needle biopsy procedures are used to diagnose prostate cancer, but current biopsy systems (standard of care control device) have been shown to underperform when compared to a new novel needle biopsy system (test device). The objectives of the study are to (1) compare tissue quality between test and control devices; (2) compare diagnostic ambiguity between the two devices; and (3) compare tissue area, length, and tortuosity from the samples with a computational pathology algorithm. Tissue analyses will be completed by pathologists blinded to the biopsy system used.

ELIGIBILITY:
Inclusion Criteria:

* Adult males with PSA density greater than or equal to 0.15
* Lesions are visible under MRI
* PIRADS score is greater than or equal to 3
* Able to and willing to provide consent

Exclusion Criteria:

* Subject has had previous local prostate therapy, focal therapy, brachytherapy, ADT, surgery, or chemotherapy for prostate cancer
* History of dementia, cognitive impairment, or deep vein thrombosis (DVT)
* Is a prisoner currently or has a history of incarceration
* Unable to understand English
* Has metastatic prostate cancer or a tumor stage of T2c, T3, or T4
* Has concurrent malignancies
* Is positive for HIV, HBV, and/or HCV infection
* Has low-performance status

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males, since only males have a prostate.
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Atypical Small Acinar Proliferation | From enrollment to end of treatment at 1 day
  Presence of suspicious prostate gland cells that appear cancerous but are not definitive enough to diagnose cancer
Gleason Score | From enrollment to end of treatment at 1 day
  Pathologist scores the biopsy sample for the percentage of samples with a Gleason score of 7, 8, 9 or 10.
Tissue area and length | From treatment to end of pathology review at 2 days
  The amount of tissue retrieved by either biopsy systems-- area and length-- will be measured using computational pathology and compared
Tissue toruosity | From treatment to end of pathology review at 2 days
  Tortuosity will be ranked from Tier 1 (high quality) to Tier 4 (low quality) using the computational pathology algorithm.

SECONDARY OUTCOMES:
Standard Pathology versus Computational Pathology Results | From treatment to end of pathology review at 2 days
  Tissue samples will be analyzed by standard pathology techniques and computational pathology and differences in values of diagnosis, Gleason score, percent tumor volume, presence of cribiform glands, and perineural invasion compared

CONTACTS AND LOCATIONS:
Overall Officials: Ted Belleza, Study Director — Uro-1 Medical

IPD SHARING:
Plan to Share IPD: No